CLINICAL TRIAL: NCT07089654
Title: Development and Evaluation of a Psychomotor Rehabilitation Nursing Plan for the Older Adults With Mild Cognitive Impairment to Promote Cognitive Health
Brief Title: Evaluation of a PMT Rehabilitation Nursing Plan for the Older Adults With MCI to Promote Cognitive Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinzhou Medical University (Other)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Wang Ying, Lecture, Jinzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JZMULL2025230; USM/JEPeM/PP/24090806 (Other: Human Research Ethics Committee USM)
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: PMT rehabilitation nursing plan
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This experimental method will be used in Quasi-Experimental Design (Non-randomized controlled trial) with experiment and control groups for comparison. Ethics consideration on older adults which would psychologically and emotionally impact in case not selected for experimental group. This research will be carried out in Liaoning Province of China. The rehabilitation nursing intervention will be carried out for older adults with MCI admitted in two China elderly care institutions which the name is Jinzhou Pension Comprehensive Service Center (JPCSC) and Jinzhou Rehabilitation Hospital (JRH). Because of ethical consideration on older adults for logistical and economical wise, easy to travel, practical, less budget. So the experimenatl group is JRH, and the control group is JPCSC. Purposive sampling, whereby older adults with MCI will be selected and invited to participate the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A PMT rehabilitation nursing plan (Experimental): Older adults will be engaged in a 12-week PMT rehabilitation nursing plan involving 2 phases of relaxation and breathing exercises, face exercises, hand exercises and mind exercises to promote cognitive health.
  Interventions: Behavioral: A PMT rehabilitation nursing plan
- General rehabilitation nursing (Other): The control group will be given a standard health education on cognitive health.
  Interventions: Behavioral: General rehabilitation nursing

INTERVENTIONS:
Behavioral: A PMT rehabilitation nursing plan — Older adults will be engaged in a 12-week PMT rehabilitation nursing plan involving 2 phases of relaxation and breathing exercises, face exercises, hand exercises and mind exercises to promote cognitive health. Phase 1 (Weeks 1-6): Includes relaxation and breathing exercises (10 minutes), facial exercises (10 minutes), bead maze activities (10 minutes), geometric shape puzzles (10 minutes), and finger exercises (20 minutes). Phase 2 (Weeks 7-12): Includes relaxation and breathing exercises (10 minutes), Tai Chi ball exercises (10 minutes), screw and nut assembly activities (10 minutes), tangram puzzles (10 minutes), and upper limb music exercises (20 minutes). The experimental group will be given interventions, twice a week every Tuesday and Thursday 9-10 am along with the study intervention.
  Arms: A PMT rehabilitation nursing plan
Behavioral: General rehabilitation nursing — The control group will be given a standard health education on cognitive health.
  Arms: General rehabilitation nursing

SUMMARY:
With the aging of the population, the number of older adults with mild cognitive impairment (MCI) has increased year by year, which has caused serious social and family burdens. At present, the existing drug treatment effect is limited. Studies show the application value of non-drug treatment in the older adults with mild cognitive impairment. Psychomotor Therapy (PMT) is now widely used in European countries and has formed an independent scientific system. Therefore, this topic pays attention to older adults with mild cognitive impairment, intending to promote cognitive stimulation, using PMT methods to build a rehabilitation nursing plan. Relying on older adults care institutions, older adults with mild cognitive impairment in a certain period were divided into a control group (CG) and an experimental group (EG). Older adults will be engaged in a 12-week PMT rehabilitation nursing plan involving relaxation and breathing exercises, face exercises, hand exercises, and mind exercises to promote cognitive health. SPSS 28.0 software was used to analyze data. The comparison of scores of various scales are based on paired t-test statistical methods. The P value <0.05 will be considered to indicate statistically significant with 95% confidence interval (CI). The rehabilitation effect of the two groups was evaluated according to cognitive assessments (Montreal Cognitive Assessment, MoCA), psychological assessment (Positive and Negative Syndrome Scale, PANSS), and emotional assessment (Hamilton Depression Rating Scale, HAMD-17; Hamilton Anxiety Rating Scale, HAMA-14) . The expected findings of this study may be useful for cognitive rehabilitation plans for the elderly in care institutions, rehabilitation hospitals, communities, and families.

DETAILED DESCRIPTION:
Introduction Research background In the wake of demographic shifts, China is experiencing the profound effects of an aging population. In 2022, China's population aged 65 and over was estimated to be 196 million, accounting for nearly 13.7% of the total population. With the change in population structure, China faces unprecedented challenges in health care, social welfare, and economic sustainability, which has a profound impact on the aging of the population, and cognitive impairment has become the most prominent problem in an aging society. Studies have shown that the overall prevalence of cognitive impairment in people aged 60 years and above in China is estimated to be 6% (95% CI: 5.8% ～ 6.3%), which increases the pressure on families, caregivers, and the healthcare system, and poses economic challenges to the country.

Similarly, population aging is a general trend around the world. According to the United Nations, by 2050, 1/6 of people in the world will be over 65 years old, compared to 1/11 in 2019. As the number of elderly people increases year by year, the prevalence of cognitive impairment in older adults is also increasing. It is reported that about 5-10% of people over 60 years old in the world suffer from dementia. Dementia is a disease characterized by cognitive decline with memory loss and impaired judgment. It not only affects the quality of life but also puts tremendous pressure on the world's healthcare systems and social support systems. Effective intervention measures are urgently needed to address this public health problem.

Mild Cognitive Impairment (MCI) refers to the prodromal stage of dementia that generally does not severely affect daily functioning, associated with an increased risk for Alzheimer's disease and other dementia. The clinical manifestations of MCI mainly include the decline of memory, language function, attention, executive function, visual-spatial structural function, and calculation ability, as well as sensory impairment and thinking disorder. While not all individuals with MCI will develop dementia. Studies have shown that MCI patients have a much higher risk of developing dementia than people with normal cognition. Early identification and intervention of MCI patients can slow or prevent the progression of dementia, thereby reducing the personal, social, and economic burden of dementia.

In recent years, there has been a large amount of literature in China that explores various aspects of dementia, including risk factors, biomarkers, diagnostic criteria, and intervention strategies. However, there are still some limitations for MCI. The diagnostic criteria and assessment tools for MCI in the Chinese population are still not unified, resulting in differences in prevalence estimates and diagnostic methods in different studies. In addition, there are insufficient longitudinal studies on the progression of MCI to dementia in older adults in China, which limits our exploration of the trajectory of the disease. Similarly, there is still no consensus on the heterogeneity of the MCI population, inconsistent diagnostic criteria, and the best treatment methods. Furthermore, the translation of research findings into clinical practice remains a significant bottleneck, with few evidence-based interventions available for preventing or delaying the onset of dementia among individuals with MCI.

Alzheimer's Disease International has advocated for and funded several studies, including some investigating the effectiveness of pharmacological and non-pharmacological interventions for early dementia. There is a great deal of ongoing research into pharmacological treatments, but traditionally, less research has been done into non-pharmacological treatments. Interventions can be broadly divided into those aimed at modifying the course of the disease, those targeting the cause of the disease, and those controlling the manifestations of the disease. PMT is often considered to fall into the last category because they may help slow cognitive decline, address symptoms related to psychosocially challenging behaviors, and improve quality of life.

Problem statement At present, there is a lot of discussion on MCI and dementia prevention. In addition to drug treatment, non-drug treatment is also a hot issue, such as music therapy, transcranial magnetic stimulation (TMS), light therapy (phototherapy), electrotherapy, acupuncture therapy, Taijiquan, Baduanjin, hyperbaric oxygen therapy (HBOT), memory therapy, etc. At present, most of the non-drug treatments target a relatively single cognitive domain, and it is difficult to solve the decline of multiple cognitive domains with one therapy. It still needs more research and discussion.

PMT is not a traditional biological model, but a kind of rehabilitation therapy under the biological-psychological-social model, which focuses on the concept of integrity. It is not focused on motor functions, but on motor skills in relationships, and is related to emotional, sensory, and cognitive functions. By mobilizing the initiative of dementia patients, stimulating their own weakened function, and assisting with personalized PMT treatment plans, a better effect of rehabilitation nursing treatment is achieved. Few published literature has applied PMT theory to the rehabilitation treatment of older adults with MCI, and the intervention plans are not uniform. At present, PMT therapy just started in China. Is it effective for older adults with MCI in China? Which group is it applicable to? Do older adults and their families accept them? There are few studies on it.

The purpose of this study is to develop a PMT rehabilitation nursing plan and evaluate the effectiveness of the rehabilitation nursing plan in older adults with MCI. The findings of this study may be useful for future studies and provide useful reference for nursing care homes, rehabilitation hospitals, communities, and families.

Research Question(s)

1. Is the PMT rehabilitation nursing plan effective in promoting cognitive health for older adults with MCI?
2. How does the PMT rehabilitation nursing plan affect the cognitive health in older adults?

Objective General: This study aimed to develop a psychomotor rehabilitation nursing plan and elucidate the effect of the PMT rehabilitation nursing plan among older adults with mild cognitive impairment in promoting cognitive function.

Specific:

1. To develop the psychomotor therapy (PMT) rehabilitation nursing plan through Delphi method for older adults with mild cognitive impairment (MCI) in promoting cognitive function.
2. To validate the psychomotor therapy (PMT) rehabilitation nursing plan for older adults with mild cognitive impairment (MCI) through content and face validation.
3. To evaluate the effectiveness of the psychomotor rehabilitation nursing plan in enhancing cognitive function among older adults with mild cognitive impairment.

Methodology Description of methodology

1. Research design: Quasi-Experimental Design (Non-randomized controlled trial) with experiment and control groups for comparison. Because of ethical considerations on older adults for logistical and economical wise, easy to travel, practical, less budget. Similar studies involving rehabilitation or behavioural interventions in real-world settings have widely used quasi-experimental designs. Studies by MA Handley and AD Harris demonstrated reliable outcomes using this approach.
2. Study area: Liaoning Province, China.
3. Study population i) Reference population: Older adults living in Liaoning. ii) Source population / sampling pool: Elderly care institutions and rehabilitation centers, Liaoning Province.

iii) Target population: Jinzhou Comprehensive Elderly Care Institution and Rehabilitation Center, Liaoning Province.

iv) Sampling frame: List of members from the two elderly care institution and rehabilitation center; Jinzhou Pension Comprehensive Service Center (JPCSC), and Jinzhou Rehabilitation Hospital (JRH), Liaoning Province.

The data collection form was created by the researcher to record general information about older adults, such as age, gender, education level, family history of dementia, marital status, personal annual income, chronic disease. It will take no more than 5 minutes. Then, It will conduct questionnaire surveys before the intervention (baseline) and after the intervention (12 weeks). The questionnaires involved include Montreal Cognitive Assessment (MoCA), which has 11 questions and takes about 10 minutes; Positive and Negative Syndrome Scale (PANSS), which has 30 questions and takes about 20 minutes; Hamilton Anxiety Rating Scale (HAMA-14), which has 14 questions and takes about 10 minutes; Hamilton Depression Rating Scale (HAMD-17), which has 17 questions and takes about 15 minutes. All questionnaires will take no more than 60 minutes. Due to ethical issues, the names of the elderly participating in this study are only used for data collection, and their identity information will not be disclosed.

Data entry and analysis will be performed using SPSS 28.0 software. Descriptive statistics will be used to summarize the general information of older adults. Numerical data will be presented as mean (SD) or median (IQR) based on their normality distribution. Categorical data will be presented as frequency (%). The comparison of scores of various scales are based on paired t-test statistical methods. The P value <0.05 will be considered to indicate statistically significant with 95% confidence interval (CI).

ELIGIBILITY:
Inclusion Criteria:

1. Older adults are aged 50 years and above.
2. Subjective cognitive complaints from the individual or caregiver.
3. Screening for MCI using the Mini-Cog scores between 0-2 ( SN Abayomi, 2024).
4. Basic language communication, listening, speaking, and understanding skills.
5. Ability to provide informed consent.

Exclusion Criteria:

1. Diagnosed with severe psychiatric conditions (e.g., schizophrenia, major depressive disorder).
2. It is at the end stage of important functional organ diseases, such as malignant tumors, cardiac failure, etc.
3. Limb dysfunction.
4. Diagnosed with dementia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive assessment | From baseline (pre-intervention) to the end of the intervention (after-intervention) at 12 weeks.
  The cognitive status of older adults will be assessed by the Montreal Cognitive Assessment (MoCA) scale. Developed by Nasreddine et al. in Canada with reference to the MMSE, the MoCA evaluates multiple cognitive domains, including attention, executive function, memory, language, visuospatial skills, abstract thinking, calculation, and orientation, making it suitable for a comprehensive assessment of various types of cognitive impairment.
  The Montreal Cognitive Assessment (MoCA) scale has a minimum score of 0 and a maximum score of 30, with higher scores indicating better cognitive function (e.g., scores near 30 reflect normal cognition), while lower scores suggest greater cognitive impairment. In Western countries, a cutoff score of 26 is commonly used to identify MCI.The results below 26 typically warrant clinical concern, though individuals with ≤12 years of education often receive a +1 point adjustment to their total score.

SECONDARY OUTCOMES:
Psychological assessment | From baseline (pre-intervention) to the end of the intervention (after-intervention) at 12 weeks.
  The psychological of older adults will be assessed by the Positive and Negative Syndrome Scale (PANSS), including the positive scale (7 items, 7~49 points), the general psychopathology scale (16 items, 16~112 points), and the negative scale (7 items, 7~49 points). The higher the score is, the worse the rehabilitation.
  The Positive and Negative Syndrome Scale (PANSS) has a minimum score of 30 (indicating absence of all measured symptoms) and a maximum score of 210 (representing severe pathology across all items). Higher PANSS scores indicate worse clinical outcomes, reflecting greater severity of psychotic symptoms-where elevated scores correlate with more pronounced positive symptoms (e.g., delusions/hallucinations), negative symptoms (e.g., social withdrawal), and general psychopathology (e.g., anxiety/impulsivity). Scores above 60 typically suggest clinically significant psychosis, with severe impairment often indicated by scores exceeding 120.
Emotional assessment | From baseline (pre-intervention) to the end of the intervention (after-intervention) at 12 weeks.
  The emotional assessment will be assessed by the Hamilton Depression Rating Scale (HAMD-17), which is among the most widely used scales for evaluating emotional status. HAMD-17 covers despair, somatization symptoms, sleep disorders, and anxiety. The Hamilton Depression Rating Scale (HAMD-17) has a minimum score of 0 (indicating no depressive symptoms) and a theoretical maximum score of 52 (though practical maxima rarely exceed 50 due to scoring constraints), with higher scores representing worse clinical outcomes-specifically greater severity of depression symptoms such as low mood, guilt, insomnia, psychomotor retardation, and suicidal ideation, where scores ≥8 suggest mild depression, ≥17 indicate moderate depression, and ≥23 reflect severe depression.
  The 2025 Expert Consensus on Neuropsychological Assessment of Mild Cognitive Impairment recommends the use of these scales, as they effectively identify and quantify depressive and anxiety symptoms in patients with MCI.
Emotional assessment | From baseline (pre-intervention) to the end of the intervention (after-intervention) at 12 weeks.
  The emotional assessment will be assessed by the Hamilton Anxiety Rating Scale (HAMA-14), which are among the most widely used scales for evaluating emotional status. The Hamilton Anxiety Rating Scale (HAMA-14) ranges from a minimum score of 0 (indicating no anxiety symptoms) to a maximum score of 56 (reflecting the most severe anxiety across all items), with higher scores signifying worse clinical outcomes-specifically greater severity of anxiety-related symptoms such as tension, fears, insomnia, and autonomic hyperactivity, where scores ≥14 typically indicate clinically significant anxiety warranting intervention, and scores >25 suggest severe impairment.
  The 2025 Expert Consensus on Neuropsychological Assessment of Mild Cognitive Impairment recommends the use of these scales, as they effectively identify and quantify depressive and anxiety symptoms in patients with MCI.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Ying Lecture Wang Ying, Master, Principal Investigator — Jinzhou Medical University / Universiti Sains Malaysia
Locations (2):
- China (2):
  - Jinzhou Pension Comprehensive Service Center, Jinzhou, Liaoning
  - Jinzhou Rehabilitation Hospital, Jinzhou, Liaoning

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlie the primary and secondary outcomes reported in publications will be shared. Data will be available upon reasonable request from 6 months after publication. Data sharing will occur through direct collaboration with the principal investigator. Interested researchers must contact wangy@jzmu.edu.cn with a scientifically justified proposal. Data sharing complies with China's Personal Information Protection Law (PIPL). International requests require approval from the local data oversight committee and sign a data use agreement.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Kwag E, Stuckenschneider T, Schneider S, Abeln V. The effect of a psychomotor intervention on electroencephalography and neuropsychological performances in older adults with and without mild cognitive impairment. Psychogeriatrics. 2021 Jul;21(4):528-539. doi: 10.1111/psyg.12702. Epub 2021 May 7. PMID 33960574
- [Background] Pereira C, Rosado H, Cruz-Ferreira A, Marmeleira J. Effects of a 10-week multimodal exercise program on physical and cognitive function of nursing home residents: a psychomotor intervention pilot study. Aging Clin Exp Res. 2018 May;30(5):471-479. doi: 10.1007/s40520-017-0803-y. Epub 2017 Aug 3. PMID 28776280
- [Background] Aziz NA, Subramaniam P, Ghazali SE, Mustafa WA. The impact of cognitive intervention on the cognition of adults over 50 with mild cognitive impairment (MCI) in Asia: A systematic review. IIUM Medical Journal Malaysia. 2022 Apr 1;21(2). doi: 10.31436/imjm.v21i2.1837
- [Background] Bruderer-Hofstetter M, Sikkes SAM, Munzer T, Niedermann K. Development of a model on factors affecting instrumental activities of daily living in people with mild cognitive impairment - a Delphi study. BMC Neurol. 2020 Jul 1;20(1):264. doi: 10.1186/s12883-020-01843-9. PMID 32611388
- [Background] Feng Z, Wu B. Embracing Challenges for Population Aging in China: Building Scientific Evidence to Inform Long-Term Care Policymaking and Practice. J Aging Soc Policy. 2023 Sep 3;35(5):543-553. doi: 10.1080/08959420.2023.2217979. Epub 2023 May 30. PMID 37249513
- [Background] Biazus-Sehn LF, Schuch FB, Firth J, Stigger FS. Effects of physical exercise on cognitive function of older adults with mild cognitive impairment: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2020 Jul-Aug;89:104048. doi: 10.1016/j.archger.2020.104048. Epub 2020 May 12. PMID 32460123
- See also: Alzheimer's Disease International. World Alzheimer Report 2021: Journey through the diagnosis of dementia. — https://www.alzint.org/resource/world-alzheimer-report-2021/
- See also: Alzheimer's Disease International. World Alzheimer Report 2011: The benefits of early diagnosis and intervention. — https://www.alzint.org/resource/world-alzheimer-report-2011/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT07089654/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT07089654/ICF_001.pdf